CLINICAL TRIAL: NCT05210764
Title: General Anesthetics-related Changes in Prefrontal EEG During Pediatric Surgical Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Other Study IDs: 2022-01-08
Record Dates: First submitted 2022-01-09; First posted 2022-01-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: General Anesthetic; Electroencephalogram
Keywords: general anesthetic; electroencephalogram
MeSH Terms: interventions — Propofol; Sevoflurane; Esketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- propofol: General anesthesia is induced and maintained mainly with propofol.
  Interventions: Drug: propofol
- sevoflurane: General anesthesia is induced and maintained mainly with sevoflurane.
  Interventions: Drug: sevoflurane
- ketamine: General anesthesia is induced mainly with S-ketamine and maintained mainly with propofol.
  Interventions: Drug: S-ketamine

INTERVENTIONS:
Drug: propofol — General anesthesia is induced and maintained mainly with propofol.
  Other Names: Propofol anesthesia group
  Groups: propofol
Drug: sevoflurane — General anesthesia is induced and maintained mainly with sevoflurane.
  Other Names: Sevoflurane anesthesia group
  Groups: sevoflurane
Drug: S-ketamine — General anesthesia is induced mainly with S-ketamine and maintained mainly with propofol.
  Other Names: S-ketamine anesthesia group
  Groups: ketamine

SUMMARY:
The change profiles of indices derived from pEEG such as phase-amplitude coupling and bicoherence based on individual general anesthetics in children have not been examined in previous literature. Whether those indices have the abilities to predict individual drug-related anesthesia depth in children need to be explored.

DETAILED DESCRIPTION:
The need to maintain a proper depth of general anesthesia during pediatric surgery is an important aspect of anesthesiology. An inappropriate anesthesia depth increases the risk of intraoperative awareness or delay in recovery in children undergoing surgery. Current modalities for anesthesia depth monitoring showed limited accuracy in children. The electroencephalogram (EEG) can be analyzed in its raw form for characteristic drug-induced patterns of change or summarized using mathematical parameters as a processed electroencephalogram (pEEG). The change profiles of indices derived from pEEG such as phase-amplitude coupling and bicoherence based on individual general anesthetics in children have not been examined in previous literature. Whether those indices have the abilities to predict individual drug-related anesthesia depth in children need to be explored.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 0-18 years, American Society of Anesthesiologists Physical Status I-II, scheduled for elective surgery in Peking University First Hospital.

Exclusion Criteria:

* Preterm patients;
* Height and weight not within the standard ranges for respective ages;
* Surgery for head or heart;
* Patients with muscular, neurologic or psychiatric diseases;
* Patients with Congenital anomaly or hereditary diseases;
* Patients with medication abuse;
* Allergy to medication including propofol, sevoflurane, and ketamine;
* Allergy to beans;
* Refusal to participate the study by guardians.

Ages: 1 Minute to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients aged 0-18 years, American Society of Anesthesiologists Physical Status I-II, scheduled for elective surgery in Peking University First Hospital
Sampling Method: Non-Probability Sample
Enrollment: 366 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
phase-amplitude coupling | induction, maintenance, and recovery of anesthesia
  phase-amplitude coupling
bicoherence | induction and maintenance, and recovery of anesthesia
  bicoherence
spectral analysis | induction and maintenance, and recovery of anesthesia
  spectral analysis
entropy indices | induction and maintenance, and recovery of anesthesia
  entropy indices

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No